CLINICAL TRIAL: NCT04278950
Title: Povidone-Iodine Rinses as an Adjuvant Therapy Post-Operatively: A Double-Blind Randomized Controlled Trial
Brief Title: Povidone-Iodine Rinses as an Adjuvant Therapy Post-Operatively
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Clinical Professor, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H19-02292
Record Dates: First submitted 2020-01-28; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Betadine; Poviodine Iodine; CRS; Biofilm; Postoperative
MeSH Terms: conditions — Disease | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poviodine Iodine Solution (Active Comparator): Patients will be randomized into this arm will be provided with 0.10% PVP-I (0.01% available iodine). Patients will be instructed to dilute 2.5mL of the betadine (unmarked bottles) into a 240mL bottle of saline and rinse once per day.
  Interventions: Drug: Povidone-Iodine
- Placebo Poviodine Iodine Solution (Placebo Comparator): Patients will be randomized into this arm will be provided with a placebo PVP-I solution. Patients will be instructed to dilute 2.5mL of the placebo PVP-I (unmarked bottles) into a 240mL bottle of saline and rinse once per day.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Povidone-Iodine — For the PVP-I group, the final concentration of available iodine in the solution will be 0.01%, (from diluting 10% PVP-I solution), as previously demonstrated to be below ciliotoxic levels of 1.25% and greater than 0.01% which is the lower limit of active potency.
  Other Names: Betadine
  Arms: Poviodine Iodine Solution
Drug: Placebos — The placebo will be 2.5mL of saline with brown food coloring.
  Arms: Placebo Poviodine Iodine Solution

SUMMARY:
Povidone Iodine solution is a nasal antiseptic. Its application has been shown to be clinically safe, tolerable and effective against bacteria and fungi associated with chronic rhinosinusitis.

The purpose of this study is determining the effectiveness of PVP-I in comparison to a placebo for post-operative refractory CRS patients in a randomized controlled trial.

DETAILED DESCRIPTION:
Background and scientific rationale Chronic rhinosinusitis (CRS) is an inflammatory condition of the paranasal sinuses affecting millions of patients, resulting in billions of dollars being spent annually in associated health care costs. Biofilm has been implicated in chronic rhinosinusitis recalcitrant to appropriate medical therapy and well-executed endoscopic sinus surgery. The presence of biofilm results in patients having worse postoperative symptoms, recurrent infections, and persistent inflammation. Biofilms are bacterial or fungi communities surrounded by an extracellular polysaccharide matrix, which facilitates attachment to mucosa, survival, protection and proliferation. This configuration allows for resistance to innate host defenses and resistance to antibiotic therapy.

Iodine bound to the synthetic carrier polymer povidone (PVP-I), has been used in wound care for several decades. The microbial activity of iodine has been thought to be facilitated through several oxidative mechanisms of action and has been shown to be effective against a wide variety of pathogens. These mechanisms include inhibition of vital bacterial cellular mechanisms, denaturation of enzymes in the respiratory chain, and oxidation of key structures in cell membranes. Previously, PVP-I-containing dressings have demonstrated complete destruction of biofilm bacteria. As well, using PVP-I as a gargle has shown bactericidal activity against methicillin-resistant Staphylococcus aureus (MRSA), Pseudomonas aeruginosa, Enterococcus faecium, among others, more so than other antimicrobials.

Use of antibiotics immediately after surgery, saline irrigation, and debridement in the office are relatively consistent post-surgical procedures for CRS patients. However, resistance to topical antibiotics such as mupirocin, fusidic acid, and gentamicin has been demonstrated in recent years. Furthermore, out of a survey of 265 otolaryngologists, it has been found that most physicians (86.8%) prescribe antibiotics following surgery, with the majority (63.9%) only taking cultures on occasion and therefore using broad-spectrum antibiotics despite issues of overuse. In contrast, resistance to PVP-I has not been documented to date and is therefore an attractive alternative in post-surgical management of CRS patients.

There is a paucity of published data on the use of iodine after sinus surgery to treat biofilm.The purpose of this study is determining the effectiveness of PVP-I in comparison to a placebo for post-operative refractory CRS patients in a randomized controlled trial.

Primary Objective:

To determine if PVP-I rinses will reduce the need for antibiotics post-FESS. The need for antibiotics will be determined by an increase in the discharge score component of the Modified Lund-Kennedy score, and/or positive Culture and Sensitivity testing.

Secondary Objective:

To assess SNOT-22 scores as well as culture and sensitivity testing which will be collected at follow-up appointments.

Baseline Evaluation

The following information will be obtained from each participant

Demographic data:

Age Gender Smoking status

Clinical data:

MLK endoscopic scores, Sinus culture and sensitivity, Blood work for inflammatory markers, Thyroid Stimulating Hormone levels, Saccharin test, Sniffin' Sticks smell test and SNOT-22 quality of life questionnaire.

Conduct of Study:

All patients undergoing primary functional endoscopic sinus surgery (FESS) at St. Paul's Hospital or False Creek Surgical Centre will be included. Patients will be randomized to receive either a placebo or 0.10% PVP-I (0.01% available iodine). Patients will be instructed to dilute 2.5mL of either the placebo or the betadine (unmarked bottles) into a 240mL bottle of saline and rinse once per day. Both groups of patients will be concurrently using the standard of care rinses as well (Pulmicort, if necessary).

For the PVP-I group, the final concentration of available iodine in the solution will be 0.01%, (from diluting 10% PVP-I solution), as previously demonstrated to be below ciliotoxic levels of 1.25% and greater than 0.01% which is the lower limit of active potency.

Should a patient develop symptoms of infection post-surgery, they will be instructed to contact the PI (Dr. Javer) or a member of his research staff. At this point they will be instructed to come for a follow-up appointment for assessment and determination of their MLK score and/or Culture and Sensitivity Testing. If they start antibiotics they will be removed from the study, and this will be indicated by censoring in the survival analysis.

Patients who do not subjectively feel unwell will come for the indicated follow-up appointments for objective and subjective assessment of their sinuses and nasal mucosa.

Management of Patient Care:

Patients have the right to withdraw from the study at any time. Patients who experience signs and symptoms of hypersensitivity to iodine, burning, itching, pain redness, tiredness, nausea or vomiting will be asked to stop the rinses immediately. The reaction will be noted and the code will be broken so that a discussion can occur between the physician and the patient regarding the use of iodine with the nasal rinses. Patients who meet any of the exclusion criteria that were not noted at the beginning of the study will be removed from this study and the physician will discuss the future management options with the patient.

Drug:

Povidone Iodine (PVP-I)

Dosing and Administration

PVP-I is provided in the form of a liquid at a concentration of 10% (1% available iodine). 2.5 mL of PVP-I will be diluted into 240 mL of saline solution. The final concentration of available iodine in the solution would be 0.01%.

Dose Schedule:

Patient will dilute 2.5 mL of 10% iodine or placebo into a 240 mL rinse bottle once a day. Both groups of patients will be concurrently using the standard of care rinses, Pulmicort, if necessary.

Duration of therapy:

The patient will administer the PVP-I or Saline rinse for 6 months

Side effects:

The literature has some isolated reports of adverse reactions to iodine administration to include burning, swelling, and pain. No documented episode of anaphylaxis due to iodine has been identified in the literature. There are reports of TSH suppression with excessive mouth gargles with iodine, however, this is quickly reverses upon cessation of use.

Sample Size:

In order to ascertain the appropriate amount of participants for a survival analysis that is sufficiently powered at 80%, the investigators will aim to complete a proof-of-concept study with 100 participant's total, 50 in each arm.

Analysis:

A survival analysis will be undertaken, with the event of interest being presence of infection in the sinuses. An 'event' will be considered a patient's need for antibiotics either by an increase in the discharge component of their MLK score and/or positive Culture and Sensitivity Testing. Time-to-event will be the duration between surgery and the point at which the patient will be removed from the study. The study period will be 6 months.

Safety Monitoring

Patients who experience signs and symptoms of iodine reaction will be noted and the code will be broken so that a discussion can occur between the research supervisor and the patient regarding the use of the topical iodine.

Patients can contact the office anytime if they notice any of the signs or symptoms of iodine reaction and will be seen by the research supervisor (or designate) within 24 hours.

Adverse Events (AE's)

All expected and unexpected adverse events will be recorded and graded by the research supervisor. Stable chronic conditions, which are present prior to the clinical trial entry and do not worsen, are not considered adverse events and will be accounted for in the patient's medical history.

Recording/Documentation of Adverse Events

During each patient visit, the research supervisor will ask appropriate questions and perform a physical exam to elicit any adverse events. The research supervisor will also review blood work obtained from the patient. All reportable adverse events will be recorded on appropriate case report form. The research supervisor will also write the stop date, the severity of the AE and his judgment of the AE's relationship to the study.

Serious Adverse Events (SAE's)

An SAE is defined as an AE meeting one of the following:

* Death occurring between Day 0 and 182 of the study.
* Life Threatening Event (defined as a participant at immediate risk of death at the time of the event)
* In-patient hospitalization or prolongation of existing hospitalization between Day 0 and 182 (6 months) of the study.

Results in a persistent or significant disability/incapacity In the event of SAE, the research supervisor will discuss with the patient (or next of kin) whether there is a relationship between the study and the SAE. If there is a relationship, the PI will be responsible for coordinating care for the patient until the SAE has been addressed.

Pregnancy During the Trial Patients will be responsible for determining if they are pregnant or become pregnant during the study. If patients notify the PI they are pregnant, they will be removed from the study and the medical management options will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* Undergoing FESS at St. Paul's Hospital or False Creek Surgical Centre

Exclusion Criteria:

* Patients with sinonasal tumors.
* Patients who previously used PVP-I rinses - Patients with autoimmune diseases affecting the upper airway

  * eg Systemic lupus erythematosus, Sjögren's syndrome, systemic sclerosis etc.
* Immuno-compromised patients, and patients with impairment in mucociliary function

  * (e.g., cystic fibrosis, Kartagener syndrome)
* Hypersensitivity to iodine
* History of thyroid disorders including thyroid cancer, hyperthyroidism and hypothyroidism
* Use of medications for thyroid disorders including thyroxine and carbimazole
* Pregnancy
* Patients unable to speak English.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-10 (Estimated); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-02-10 (Estimated)

PRIMARY OUTCOMES:
Modified Lund-Kennedy endoscopic scores | 6 months
  This score is based on the endoscopic assessment of polyps, edema, and discharge and are each given score 0-2. A higher score indicates a worse outcome.
Cultures and Sensitivity | 6 months
  Assess whether there is positive growth of bacteria or fungi.

SECONDARY OUTCOMES:
SNOT-22 | 6 months
  This is a standard of care form that includes 22 questions about symptoms and social/emotional consequences of your nasal disorder. You will be asked to rate your problems as they have been over the past two weeks. Patients give a score out of 110 where a higher score indicates a worse outcome.
Blood test | 6 months
  Serum IgE levels
Saccharin test | 6 months
  Test to assess nasal mucociliary clearance. Place a small amount of saccharin one cm behind the anterior aspect of the inferior turbinate. Normal mucociliary would result in saccharin being swept backwards to the nasopharynx, allowing the subject to taste the sweet saccharin.
Sniffin' Stick smell test | 6 months
  Many CRS patients have a disturbed/ reduced sense of smell. Sniffn' Sticks is a type of test to assess your sense of smell by using various scented pens. The threshold and identification tests will be performed. A score will be given out of 32 with a lower score indicating a worse outcome/sense of smell.
Blood test | 6 months
  Eosinophils levels

CONTACTS AND LOCATIONS:
Overall Officials: Amin Javer, MD, Principal Investigator — University of British Columbia and St. Paul's Hospital